CLINICAL TRIAL: NCT01299103
Title: A Prospective, Randomized, Open-Label, 3-Arm Parallel Study Comparing the Safety and Efficacy of Single Therapy Versus Double and Triple Therapy Using the Surgitron® Dual RF™ S5 With the Pellevé™ Wrinkle Treatment Handpiece and Pellevé™ Treatment Gel for the Treatment of Moderate Facial Wrinkles in Fitzpatrick Skin Types I - IV
Brief Title: Safety and Efficacy of Single Therapy Versus Double and Triple Therapy of the Pellevé™ Wrinkle Treatment System for the Treatment of Moderate Facial Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellman International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEL-10-02
Record Dates: First submitted 2011-02-04; First posted 2011-02-18 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Appearance of Facial Wrinkles
Keywords: wrinkle; rhytide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Treatment (Active Comparator): Treatment of facial wrinkle with one treatment only
  Interventions: Device: Pelleve Wrinkle Treatment System
- Double Treatment (Active Comparator): Treatment of facial wrinkle with two treatments
  Interventions: Device: Pelleve Wrinkle Treatment System
- Triple treatment (Active Comparator): Treatment of facial wrinkle with three treatments
  Interventions: Device: Pelleve Wrinkle Treatment System

INTERVENTIONS:
Device: Pelleve Wrinkle Treatment System — comparison of single vs. double and triple treatment with the Pelleve Wrinkle Treatment System

SUMMARY:
The study will enroll and treat a patients to assess improvement in the appearance of facial wrinkles.

DETAILED DESCRIPTION:
The study will enroll and treat a total of 44 subjects (23 in treatment Group A receiving a single treatment and 21 in treatment Group B receiving two treatments) with moderate facial wrinkles corresponding to a grade of 4-6 on the validated Fitzpatrick Wrinkle Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Females 35-60 years of age with Fitzpatrick Skin Color Type I-IV.
* Subjects with clinical evidence of facial wrinkles mild to moderate in severity as specified by a grade 4-6 on the Fitzpatrick Wrinkle Assessment Scale.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Willingness and ability to provide written photo consent and adherence to photography procedures (i.e., removal of jewelry and makeup).
* Willingness and ability to provide written informed consent prior to performance of any study related procedure.

Exclusion Criteria:

* Subjects who are pregnant, nursing, planning to become pregnant, and/or not using a reliable form of birth control.
* Subjects who have had prior exposure to any hyaluronic acid, or any other filler, injection for any purpose in the 12 months preceding study enrollment through the duration of the study.
* Subjects who have had prior exposure to any botulinum toxin for facial rhytids in the 6 months preceding study enrollment through the duration of the study.
* Subjects who have had a prior cosmetic procedure to improve facial rhytids (i.e., rhytidectomy, periorbital or eyelid/eyebrow surgery, brow lift, CO2/erbium laser resurfacing, Thermage/Thermacool radiofrequency treatment) within 12 months or who have visible scars that may affect evaluation of response and/or quality of photography.
* Ablative skin resurfacing on the glabellar area within the previous 6 months or during the study.
* Retinoid, microdermabrasion, or prescription level glycolic acid treatments within 3 months prior to study participation or during the study.
* Active cut, wound, or infection on the skin.
* Oral Isotretinon within the past 12 months.
* Active HSV-1.
* History of keloids or hypertrophic scarring.
* Existing or history of skin malignancy.
* Any existing skin disease.
* History of collagen or vascular disease.
* Subjects who have implantable pacemaker, automatic implantable defibrillator/ cadioversor (AICD), or any other implantable electric device.
* Subjects who have used, within 30 days, any medication that can cause dermal hypersensitivity or affect skin characteristics.
* History of autoimmune disease.
* History of any disease that inhibits pain sensation.
* History of Diabetes I or II.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the Investigator's opinion, have a history of poor cooperation, non¬compliance with medical treatment or unreliability.
* Enrollment in any active study involving the use of investigational devices or drugs.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research Institute, Chichago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Treatment: Subjects receive one treatment
- Double Treatment: Subjects receive two treatments
- Triple Treatment: Subjects receive three treatments
Period: Overall Study
Arm/Group | Single Treatment | Double Treatment | Triple Treatment
Started | 15 | 15 | 10
Completed | 15 | 13 | 8
Not Completed | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Treatment | Double Treatment | Triple Treatment | Total
Number analyzed (Participants) | 15 | 15 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (7.2) | 52 (6.5) | 53 (5.2) | 52 (6.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 10 | 40
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Fitzpatrick Wrinkle Assessment
Description: Subject photos will be evaluated using the 9-point Fitzpatrick Wrinkle Assessment Scale at all follow up visits. An improvement is noted by a decrease in the numeric Fitzpatrick Wrinkle score. The Fitzpatrick Wrinkle Assessment ranges from 1-9. Wrinkle Score between baseline and 90 days post treatment assessment. Positive values indicates an increase in score, while negative values indicate a decrease
Time Frame: change in Fitzpatrick Wrinkle Score between baseline and 90 days post treatment assessment.
Measure: Mean (Standard Deviation); unit: units on a scale, change in Fitzpatrick
Arm/Group | Single Treatment | Double Treatment | Triple Treatment
Number analyzed (Participants) | 15 | 13 | 8
units on a scale, change in Fitzpatrick | 1.0 (0.98) | 1.5 (1.9) | 1.1 (1.7)

2. Primary Outcome: Adverse Events
Description: The rate of adverse events occurring in treatment subjects will be assessed.
Time Frame: 90 days post treatment
Measure: Number; unit: number of adverse events reported
Arm/Group | Single Treatment | Double Treatment | Triple Treatment
Number analyzed (Participants) | 15 | 13 | 8
number of adverse events reported | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Single Treatment | Double Treatment | Triple Treatment
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/10
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No